Official Title: An Open-Label, Real World Study Evaluating the Long-Term Quality of Life

of Tildrakizumab in Adult Patients With Moderate to Severe Plaque Psoriasis

**Document:** Statistical Analysis Plan (SAP)

NCT number: NCT03718299

**Date:** 24-FEB-2021



#### STATISTICAL ANALYSIS PLAN

VERSION: 1.0

DATE: 24-FEB-2021

**SPONSOR:** Sun Pharma Global FZE

PROTOCOL NUMBER: TIL2018-1

**PROJECT NUMBER:** 177-11151-401

**PROTOCOL TITLE:** An Open Label, Real World Study Evaluating the Long-Term

Quality of Life of Tildrakizumab in Adult Patients with

Moderate to Severe Plaque Psoriasis

#### **ABBREVIATIONS**

AE Adverse Event
BSA Body Surface Area
CSR Clinical Study Report

dL Deciliter

DLQI Dermatology Life Quality Index eCRF Electronic Case Report Form HIV Human Immunodeficiency Virus I-NRS Itching Numeric Rating Scale

ITT Intent-to-Treat

MedDRA Medical Dictionary for Regulatory Activities

mL Milliliter

mIU Milli-International Units
P-NRS Pain Numeric Rating Scale
PASI Psoriasis Area and Severity Index

PP Per-Protocol PT Preferred Term

PGWB Physical General Well-Being

QoL Quality of Life

S-NRS Scaling Numeric Rating Scale

SAE Serious Adverse Event
SAP Statistical Analysis Plan
SD Standard Deviation
SOC System Organ Class

sPGA Static Physician's Global Assessment

TB Tuberculosis

TSQM Treatment Satisfaction Questionnaire for Medication

TEAE Treatment Emergent Adverse Event

UPT Urine Pregnancy Test

WOCBP Women of Childbearing Potential

WPAI-PSO Work Productivity and Activity Impairment scale - Psoriasis

# TABLE OF CONTENTS

| Ta | ble of | Con | tents | . 5 |
|---|---|---|---|---|
| 1. | Intr | oduc | tion | . 7 |
| 2. | Pur | pose | of the Analyses | . 7 |
| 3. | Stu | dy O | bjectives and Endpoints | . 7 |
| | 3.1 | | ectives | |
| | 3.2 | Effi | cacy Endpoints | . 7 |
| | 3.2. | .1 | Primary | . 7 |
| | 3.2. | .2 | Secondary | . 7 |
| | 3.3 | Safe | ety Endpoints | . 8 |
| 4. | Stu | dy D | esign | . 8 |
| 5. | Def | initio | ons | 10 |
| 6. | Cli | nical | evaluations | 10 |
| | 6.1 | Bod | y Surface Area (BSA) | 10 |
| | 6.2 | Stat | ic Physician's Global Assessment (sPGA) | 10 |
| | 6.3 | Pson | riasis Area Severity Index (PASI) | 10 |
| | 6.4 | Itch | Numerical Rating Scale (I-NRS) | 11 |
| | 6.5 | Pain | Numerical Rating Scale (P-NRS) | 11 |
| | 6.6 | Scal | ing Numerical Rating Scale (S-NRS) | 11 |
| | 6.7 | Psy | chological General Well-Being Index (PGWB) | 11 |
| | 6.8 | Den | matology Life Quality Index (DLQI) | 14 |
| | 6.9 | Wor | ck Productivity and Activity Impairment Scale (WPAI-PSO) | 15 |
| | 6.10 | <b>T</b> 1 | reatment Satisfaction Questionnaire for Medication (TSQM) | 16 |
| | 6.11 | | ildrakizumab Overall Satisfaction | |
| | 6.12 | Pa | atient Happiness with Psoriasis Control | 19 |
| | 6.13 | Fι | all-Body Photography (excluding face) | 19 |
| 7. | Saf | ety E | valuations | 19 |
| | 7.1 | Ådv | rerse Events | 19 |
| | 7.2 | Bloo | od Chemistries, Hematology, and Virology/HIV | 19 |
| | 7.3 | | ntiFERON-TB Gold test | |
| | 7.4 | Preg | gnancy Tests | 20 |
| | 7.5 | Phy | sical Exam | 20 |
| 8. | Stat | tistic | al Methods | 20 |
| | 8.1 | Gen | eral Considerations | 20 |
| | 8.2 | Ana | lysis Populations | 21 |
| | 8.2. | .1 | Safety Population | 21 |
| | 8.2. | .2 | Intent-to-Treat Population | 21 |
| | 8.2. | .3 | Per-Protocol Population | |
| | 8.3 | | Il Analyses and Reporting | |
| | 8.4 | | iple Size | |
| | 8.5 | | lysis Visit Windows | |
| | 8.6 | | ject Disposition | |
| | 8.7 | | eening and Baseline Assessments | |
| | 8.7. | | Demographics and Baseline Characteristics | |
| | 8.7. | .2 | Medical History | |

| | 8.7.3 | Baseline Clinical Evaluations | 23 |
|---|---|---|---|
| 8 | 0.7.0 | sing Compliance | |
| | .9 Effi | cacy Evaluation | 24 |
| Ü | 8.9.1 | Analysis of Efficacy | |
| 8 | | tatistical / Analytical Issues | |
| Ĭ | 8.10.1 | Handling of Dropouts or Missing Data | |
| | | Interim Analyses | |
| | 8.10.3 | Multicenter Studies | |
| | 8.10.4 | Multiple Comparisons / Multiplicity | |
| | 8.10.5 | Examination of Subgroups | |
| 8 | .11 S | afety Evaluation | |
| | 8.11.1 | Extent of Exposure | |
| | 8.11.2 | Adverse Events | |
| | 8.11.3 | Clinical Laboratory Tests | 28 |
| | 8.11.4 | Physical Examinations Error! Bookma | ark not defined. |
| | 8.11.5 | Vital Signs | ark not defined. |
| | 8.11.6 | Prior and/or Concomitant Medications and Procedures/ Therapies | 28 |
| | 8.11.7 | Protocol Deviation | ark not defined. |
| 9. | Change | s to Planned Protocol Analysis | 28 |

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) describes the planned statistical analyses to be performed for data from Protocol TIL2018-1, "An Open Label, Real World Study Evaluating the Long-Term Quality of Life of Tildrakizumab in Adult Patients with Moderate to Severe Plaque Psoriasis".

This SAP was created using Clinical Protocol TIL2018-1 Version 1.3 dated 02Jan2020, and the electronic Case Report Forms (eCRFs) Version 2.0 dated 02Jul2020.

#### 2. PURPOSE OF THE ANALYSES

The purpose of this SAP is to outline the planned analyses to be completed to support the Clinical Study Report (CSR) for Protocol TIL2018-1. Any post-hoc or unplanned analyses not identified in this SAP will be clearly identified in the CSR.

#### 3. STUDY OBJECTIVES AND ENDPOINTS

### 3.1 Objectives

The primary objective is to demonstrate improvement from baseline in patient quality of life (QoL) after 28 and 52 weeks of treatment with tildrakizumab, under real world conditions, as measured by Psychological General Well-Being scale (PGWB).

Secondary objectives include assessment of patient quality of life as measured by the Dermatology Life Quality Index (DLQI), work productivity and activity impairment, psoriasis symptom control, patient satisfaction, long-term efficacy, and safety.

#### 3.2 Efficacy Endpoints

#### 3.2.1 Primary

Improvement in quality of life measured by change from baseline in total PGWB score at Week 28 and Week 52

#### 3.2.2 Secondary

- 1. Improvement in quality of life measured by change from baseline in total PGWB score as well as PGWB scores for subscales in anxiety, depression, positive-well being, self-control, general health and vitality over time (weeks 4, 8, 12, 16, 40, 64)
- 2. Improvement in quality of life measured by change from baseline in DLQI over time (weeks 4, 8, 12, 16, 28, 40, 52, 64)
- 3. Proportion of subjects with DLQI score of 0 or 1 at weeks 4, 8, 12, 16, 28, 40, 52, and 64
- 4. Proportion of subjects with DLQI score <5 at weeks 4, 8, 12, 16, 28, 40, 52, and 64
- 5. Proportion of subjects with a reduction of  $\geq$  5 points in DLQI from baseline at weeks 4, 8, 12, 16, 28, 40, 52, and 64

6. Efficacy of drug as measured by change in percent affected body surface area (BSA), change in Static Physician's Global Assessment (sPGA), and/or BSAxPGA over time (weeks 4, 8, 12, 16, 28, 40, 52, 64)

- 7. Efficacy of drug as measured by Psoriasis Area Severity Index (PASI) (% of PASI improvement from baseline, absolute PASI) over time (weeks 4,16, 28, 52)
- 8. Improvement from baseline in itch, pain, and scaling using numerical rating scales over time (weeks 4, 8, 12, 16, 28, 40, 52, 64)
- 9. Proportion of patients with itch score of 0, pain score of 0, and scaling score of 0, respectively, at weeks 4, 8, 12, 16, 28, 40, 52, and 64
- 10. Improvement from baseline in work productivity measured by change in Work Productivity and Activity Impairment scale (WPAI-PSO) over time (weeks 16, 28, 40, 52, 64)
- 11. Assessment of patient satisfaction with treatment measured with Treatment Satisfaction Questionnaire for Medication (TSQM) over time (weeks 4, 8, 12, 16, 28, 40, 52, 64)
- 12. Tildrakizumab overall satisfaction over time (weeks 4, 8, 12, 16, 28, 40, 52, 64)
- 13. Patient happiness with psoriasis control over time (weeks 4, 8, 12, 16, 28, 40, 52, 64)

### 3.3 Safety Endpoints

Incidence (severity and causality) of any local and systemic adverse events (AEs).

#### 4. STUDY DESIGN

This is a Phase 4 multicenter, uncontrolled open-label study design. There will be a total of 10 study visits at Screening, Baseline, Week 4, Week 8, Week 12, Week 16, Week 28, Week 40, Week 52 and Week 64, with subjects receiving tildrakizumab injections at Week 0, Week 4, Week 16, Week 28, Week 40, and Week 52. The total study duration will be approximately 64 weeks, excluding a screening period. Approximately 60 subjects will be enrolled into the study at two sites. For an individual subject, the study duration should be approximately 64 weeks. The duration of the study as a whole will vary based upon the rate of recruitment and completion of subjects.

Sponsor: Sun Pharma Global FZE

| _ | tical Analysis Plan, v1.0<br>oject: 177-11151-401 | Sponsor: Sun Pharmaceuticals Global FZE<br>Protocol Number: TIL2018-1 |
|---|---|---|
| 5. | The Study Day is the day of the study product. The baseline assessment is defined to the color of the study product. Change from Baseline will be calcon to the color of the | d as the measurement collected at application of the study product. |
| 6. | CLINICAL EVALUATIONS | |
| 6.1 | Body Surface Area | |
| The p | percent BSA affected with psoriasis | will be estimated at each study visit. |
| 6.2 | Static Physician's Global Assessn | nent |
| | | severity of psoriasis lesions at a given time point. The re according to following classification: |
| 6.3 | Psoriasis Area Severity Index | |
| | | neasuring the severity of psoriatic lesions based on area<br>alyzes the four regions of the body (head, trunk, upper |

and lower limbs)

. A higher score

indicates more severe disease.







## 6.8 Dermatology Life Quality Index

The DLQI is a self-administered and user-friendly validated questionnaire used to measure the health-related quality of life of adult patients suffering from a skin disease. It consists of questions concerning patients' perception of the impact of skin diseases on different aspects of their health related quality of life over the last week. The items of the DLQI encompass aspects such as symptoms and feelings, daily activities, leisure, work or school, personal relationships and the side effects of treatment. Scores of individual items

Higher scores mean greater impairment of patient's QoL.



# 6.9 Work Productivity and Activity Impairment Scale

The WPAI is a validated, subject-reported quantitative assessment of the amount of absenteeism, presenteeism and daily activity impairment attributable to general health or a specific health problem. WPAI surveys were analyzed based on published algorithms to determine the following: current employment status, absenteeism , presenteeism total activity impairment , and total work productivity impairment higher scores representing greater impairment (worse outcomes).



## 6.10 Treatment Satisfaction Questionnaire for Medication

The TSQM is a general measure of treatment satisfaction with medication, suitable for use across a wide variety of medication types and illness conditions. The TSQM Version 1.4 is a reliable and valid instrument to assess patients' satisfaction with medication, providing scores on four scales – side effects, effectiveness, convenience and global satisfaction.

TSQM consists of fourteen questions. It will be computed and summarized by adding the items in each of the four domain below. This provided a transformed score between that should be

rating scale that is administered at each visit starting at Visit 3 (Week 4). Subjects indicate their overall satisfaction with the use of tildrakizumab as well as on specific areas by circling the integer

# 6.12 Patient Happiness with Psoriasis Control

The Patient Happiness with Psoriasis Control assessment is a simple, self- administered numeric rating scale that is administered at each visit.

Subjects indicate their overall happiness with psoriasis control by circling the integer that best describes their experience on an scale

### 6.13 Full-Body Photography (excluding face)

Full-body photographs will be taken on consenting subjects. Clinical photographs should be standardized using a solid color background and consistent subject positioning and lighting. Approximately views should be taken; full front, full back and four half-body views, ensuring that all non-head areas affected by psoriasis are captured. Subjects who refuse to undergo full-body photography may still be enrolled in the study. Photos are only for visual documentation of psoriasis and will not be analyzed.

### 7. SAFETY EVALUATIONS

#### 7.1 Adverse Events

An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE (also referred to as an adverse experience) can be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, without any judgment about causality. An AE can arise from any use of the drug (e.g., off-label use, use in combination with any drug) and from any route of administration, formulation, or dose, including an overdose. A treatment emergent AE (TEAE) is defined as an AE that started on or after the date of the first dose of test article.

The severity of an AE will be recorded as mild, moderate, or severe. The relationship between an AE and the test article will be classified as definitely related, probably related, possibly related, unlikely related, or not related.

### 7.2 Blood Chemistries, Hematology, and Virology/Human Immunodeficiency Virus

Blood samples for laboratory tests are to be taken prior to first administration of test article and should be performed according to standard laboratory procedures. Follow-up labs for chemistry, blood count and virology beyond screening can be done at the clinical judgment of the investigator.

### 7.3 QuantiFERON-Tuberculosis Gold test

QuantiFERON-Tuberculosis (TB) Gold test is not required at screening for subjects with a history of latent TB and ongoing treatment for latent TB or documentation of having completed appropriate treatment. Subject is to undergo chest x-ray during Screening period if result of QuantiFERON-TB Gold test is positive, or if they have history of latent TB, signs or symptoms suggestive of active TB or had recent close contact with a person with active TB.

#### 7.4 Pregnancy Tests

A serum pregnancy test must be performed on all female subjects of child-bearing potential at A urine pregnancy test (UPT) will be performed in women of childbearing potential at all visits where study article is administered.

#### 7.5 Physical Exam

A full physical exam including vital signs, height and weight will be performed at . The limited physical exam with vital signs and weight will be performed at .

#### 8. STATISTICAL METHODS

#### 8.1 General Considerations

All statistical processing will be performed using SAS® Version 9.4 or higher, unless otherwise stated. For continuous variables, descriptive statistics will include the number of subjects with non-missing data (n), mean, standard deviation (SD), median, minimum, and maximum values. For categorical variables, the number and percentage of subjects within each category will be

presented. Subject data listings will be sorted by treatment group, study site and subject number and visit, as applicable.

## 8.2 Analysis Populations

All subjects will be classified into the Intent-to-Treat (ITT), Per-Protocol (PP), and Safety populations according to the following definitions. Membership in the analysis populations will be determined prior to database lock.

### 8.2.1 Safety Population

The Safety population will include all subjects who are enrolled

## 8.2.2 Intent-to-Treat Population

The ITT population will include all subjects who are enrolled

### 8.2.3 Per-Protocol Population

The Per Protocol Population will include a subset of the ITT population who completed the study and meet the following criteria:

1. Meets all inclusion/exclusion criteria

# 8.3 Final Analyses and Reporting

Final database lock will occur after all subjects have completed the study assessment period (or discontinued early) and all subject data has been monitored. Analysis may not occur until after this SAP is approved, analysis populations have been identified and database lock.

### 8.4 Sample Size

No formal sample size calculations were performed. The sample size of 60 subjects was selected to provide adequate estimates of probable events in the population.

#### 8.5 Analysis Visit Windows

Efficacy data will be assigned to analysis visits based on its nominal scheduled visit. Early termination visit will be assigned to analysis visits as defined in the visit window tables below.

Final visit is the subject's last visit. If the subject completed the study, Week 64/Visit 10 will be the last visit; if a subject discontinued, the efficacy data for the last visit will be assigned to the analysis visit defined by the analysis visit window.



# 8.6 Subject Disposition

The number and percentage of subjects who were enrolled in the study, in each analysis population, who completed the study, who withdrew from the study and their reasons for discontinuation will be summarized.

Protocol deviations will be summarized by total deviations and by deviations type for Safety population with available data, using descriptive statistics.

### 8.7 Screening and Baseline Assessments

### 8.7.1 Demographics and Baseline Characteristics

Demographic and baseline characteristics including age, sex, ethnicity and race will be summarized by treatment group for the ITT, PP and Safety populations using descriptive statistics. Demographic data for screen failures will be summarized separately.

### 8.7.2 Medical History

Medical histories will be provided in a subject listing for the Safety population. Findings noted during the Screening and Baseline physical examinations will be recorded in the medical history.

## 8.7.3 Psoriasis Treatment History

Psoriasis treatment history will be summarized by number and percentage of subjects for each type of prior treatment and also the number and percentage of subjects with each clinical response for each treatment. A subject listing for individual psoriasis treatment history will be provided.

#### 8.7.4 Physical Examinations

Physical examination results will be included in medical history.

### 8.7.5 Vital Signs, Height, Weight and Body Mass Index

Descriptive statistics of the observed and change from Baseline values of each vital sign parameter (temperature, systolic and diastolic blood pressure, heart rate, and respiration rate) and weight will be provided for each scheduled visit. Descriptive statistics of height and body mass index will be provided at Screening/Baseline.

#### 8.7.6 Baseline Clinical Evaluations

The Screening and Baseline severity scores for sPGA will be tabulated for the ITT population. Descriptive statistics will be provided for the Screening and Baseline data of BSA, PASI, WPAI-PSO, PGWB, DLQI, I-NRS, P-NRS, S-NRS and Patient Happiness with Psoriasis control.



### 8.9 Efficacy Evaluation

## 8.9.1 Analysis of Efficacy

The efficacy analyses will be conducted on the ITT population and repeated on the PP population for selected endpoints. The Safety population will be used for the analyses of safety endpoints.

Change from Baseline for the efficacy variables will be analyzed using the t-test. The 95% 2-sided confidence intervals will be calculated.

For dichotomous response variables, the binomial exact 95% confidence interval will be presented.

For all efficacy by visit analysis, a final visit will be included. The final visit is either Week 64/Visit 10 if a subject completed the study, or the last visit before discontinuation.

#### **BSA**

The BSA will be analyzed for the following endpoint:

• Change from Baseline to Weeks 4, 8, 12, 16, 28, 40, 52 and 64, with percent Change from Baseline summarized

# **sPGA**

The sPGA will be analyzed for the following endpoint:

- Change from Baseline to Week 4, 8, 12, 16, 28, 40, 52 and 64
- The proportion of subjects with a ≥1-grade decrease from Baseline to each study visit
- The proportion of subjects with a ≥2-grade decrease from Baseline to each study visit
- The proportion of subjects categorized as 'clear' (0) or 'almost clear' (1) on the sPGA and a ≥2-grade decrease from Baseline to each study visit

#### BSA x sPGA

The product of BSA x sPGA will be analyzed for the following endpoint:

 Change from Baseline to Weeks 4, 8, 12, 16, 28, 40, 52 and 64, with percent Change from Baseline summarized

#### **PASI**

The PASI total score will be analyzed for the following endpoint:

 Change from Baseline to Weeks 4, 16, 28 and 52, with percent Change from Baseline summarized





#### I-NRS

- Change from Baseline to Weeks 4, 8, 12, 16, 28, 40, 52 and 64, with percent Change from Baseline summarized
- Proportion of patients with I-NRS of 0 at Weeks 4, 8, 12, 16, 28, 40, 52 and 64

### P-NRS

- Change from Baseline to Weeks 4, 8, 12, 16, 28, 40, 52 and 64, with percent Change from Baseline summarized
- Proportion of patients with P-NRS of 0 at Weeks 4, 8, 12, 16, 28, 40, 52 and 64

#### S-NRS

- Change from Baseline to Weeks 4, 8, 12, 16, 28, 40, 52 and 64, with percent Change from Baseline summarized
- Proportion of patients with S-NRS of 0 at Weeks 4, 8, 12, 16, 28, 40, 52 and 64

## **PGWB**

The PGWB score will be analyzed for the following endpoint:

- Change from Baseline to Weeks 4, 8, 12, 16, 28, 40, 52 and 64 in global score, with percent Change from Baseline summarized
- Change from baseline to Weeks 4, 8, 12, 16, 28, 40, 52 and 64 in each of the six sub domain, with percent Change from Baseline summarized

#### DLQI

DLQI will be analyzed for the following endpoint:

- Change from Baseline to Week 4, 8, 12, 16, 28, 40, 52 and 64 in DLQI total score, with percent Change from Baseline summarized
- The proportion of subjects with DLQI total score of 0 or 1 at Weeks 4, 8, 12, 16, 28, 40, 52 and 64
- The proportion of subjects with DLQI total score ≤5 at Weeks 4, 8, 12, 16, 28, 40, 52 and 64
- The proportion of subjects with a reduction of ≥5 points in DLQI total score from Baseline at Weeks 4, 8, 12, 16, 28, 40, 52 and 64. Subjects must have Baseline DLQI score of ≥5 to be included in this analysis.

#### WPAI-PSO

Each of the four WPAI-PSO domain scores will be analyzed for the following endpoint:

Change from Baseline to Weeks 16, 28, 40, 52 and 64.

## **TSQM**

Each of the four TSQM domain scores at Weeks 4, 8, 12, 16, 28, 40, 52 and 64



## **Tildrakizumab Overall Satisfaction**

Tildrakizumab Overall Satisfaction score in each of the four specific areas will be summarized for Weeks 4, 8, 12, 16, 28, 40, 52 and 64.

## Patient Happiness with Psoriasis Control

Patient Happiness with Psoriasis Control will be analyzed for the following endpoint:

 Change from Baseline to Weeks 4, 8, 12, 16, 28, 40, 52 and 64, with percent Change from Baseline summarized

#### 8.10 Statistical / Analytical Issues



#### 8.10.2 Interim Analyses

Interim analysis is planned to be performed after all subjects have reached Week 28. All available data up to the date when subjects complete Week 28 (or discontinue prior to completing Week 28) will be included in the interim analysis as described below. Efficacy data will be summarized for the ITT population only.

- Demographics
- PGWB score percent change from baseline at weeks 4, 8, 12, 16, 28, 40, 52, and 64
- Proportion of subjects with DLQI score of 0 or 1 at weeks 4, 8, 12, 16, 28, 40, 52, and 64
- Efficacy of drug as measured by BSA, sPGA, and BSA x sPGA at weeks 4, 8, 12, 16, 28, 40, 52, 64; Subgroup group analysis based on Baseline BMI
- PASI score absolute and percent change from Baseline at weeks 4,16, 28 and 52; Subgroup group analysis based on Baseline BMI
- Improvement from baseline in itch, pain, and scaling using numerical rating scales over time (weeks 4, 8, 12, 16, 28, 40, 52, 64)
- Proportion of subjects with itch score of 0, pain score of 0, and scaling score of 0, respectively, at weeks 4, 8, 12, 16, 28, 40, 52, and 64

- Assessment of patient satisfaction with treatment measured with Treatment Satisfaction Questionnaire for Medication (TSQM) at weeks 4, 8, 12, 16, 28, 40, 52, 64
- Tildrakizumab overall satisfaction at weeks 4, 8, 12, 16, 28, 40, 52, 64
- Patient happiness with psoriasis control at weeks 4, 8, 12, 16, 28, 40, 52, 64
- Adverse events

#### 8.10.3 Multicenter Studies

All study sites adhered to the same protocol and will have their data pooled for summary purposes.

## 8.10.4 Multiple Comparisons / Multiplicity

No multiplicity adjustment is planned in this study.

### 8.11 Safety Evaluation

#### 8.11.1 Extent of Exposure

Descriptive statistics will be used to summarize the treatment duration, total number of injections, and the percent of expected injections taken for the Safety, ITT and PP populations.

#### 8.11.2 Adverse Events

AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). Verbatim terms will be mapped into a MedDRA system organ class (SOC) and preferred term (PT). For all AE summaries, if a subject has more than one AE within a PT, the subject is counted once in that preferred term. If a subject has more than one AE within a SOC, the subject is similarly counted once in that SOC.

The number and percentage of unique subjects reporting each TEAE will be summarized by SOC and PT. The number and percent of unique subjects reporting each treatment-emergent AE will also be summarized by SOC, PT, and maximum severity (mild, moderate, severe) and closest relationship to test article (not related, unlikely, possibly, probably, definitely).

SAEs, if any, will be summarized by SOC, PT and treatment group.

AE listing will be provided and CTCAE grade will be included.

### 8.11.3 Clinical Laboratory Tests

All laboratory data (hematology, chemistry, and serum) will be listed and reported in the units received by the laboratory. Descriptive statistics will be provided for Screening visit.

A listing of UPT results will also be provided.

Result from QuantiFERON-TB Gold test and chest x-ray during Screening period if result of QuantiFERON-TB Gold test is positive will also be provided in a subject listing.

## 8.11.4 Prior and/or Concomitant Medications and Procedures/ Therapies

Prior and/or concomitant medications and concurrent therapies/procedures will be provided in subject listings.

#### 9. CHANGES TO PLANNED PROTOCOL ANALYSIS

None.